CLINICAL TRIAL: NCT06970678
Title: Efficacy of Dexmedetomidine Infusion Combined With Paragastric Neural Block in Enhancing Postoperative Recovery Following Laparoscopic Sleeve Gastrectomy
Brief Title: Combining Dexmedetomidine Infusion and Paragastric Autonomic Neural Block to Enhance Postoperative Recovery in Patients Undergoing Laparoscopic Sleeve Gastrectomy
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16/463
Record Dates: First submitted 2025-04-15; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Laparoscopic Sleeve Gastrectomy (LSG)
Keywords: dexmedetomidine infusion; laparoscopic sleeve gastrectomy (LSG); paragastric neural block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients receiving Dexmedetomidine infusion plus PGANB (Experimental): Patients will receive intravenous loading dose of dexmedetomidine at 0.5 μg/kg ideal body weight (concentration 2 μg/ml) over 15 minutes prior to anesthesia induction, followed by 10 ml of 0.9% sodium chloride over 60 seconds during anesthetic induction. Post-intubation, Dexmedetomidine will be maintained at 0.5 μg/kg/h ideal body weight via a syringe pump until trocar removal.
  Paragastric autonomic neural block (PGANB) will be administered using a 25-gauge needle attached to a venous catheter extension, introduced through the left 12 mm port. Infiltration of 20 mL undiluted 0.5% bupivacaine will be performed at six levels in the fatty tissue of the paragastric area, including the lesser omentum, vagus nerve, esophagogastric junction, proximal stomach, mid-stomach, distal antrum, hepatic artery, and left gastric artery, with the needle cap removed under direct vision throughout the procedure.
  Interventions: Drug: Dexmedetomidine infusion; Procedure: paragastric autonomic neural block

INTERVENTIONS:
Drug: Dexmedetomidine infusion — Patients will receive intravenous loading dose of dexmedetomidine at 0.5 μg/kg ideal body weight (concentration 2 μg/ml) over 15 minutes prior to anesthesia induction, followed by 10 ml of 0.9% sodium chloride over 60 seconds during anesthetic induction. Post-intubation, Dexmedetomidine will be maintained at 0.5 μg/kg/h ideal body weight via a syringe pump until trocar removal.
Procedure: paragastric autonomic neural block — Paragastric autonomic neural block (PGANB) will be administered using a 25-gauge needle attached to a venous catheter extension, introduced through the left 12 mm port. Infiltration of 20 mL undiluted 0.5% bupivacaine will be performed at six levels in the fatty tissue of the paragastric area, including the lesser omentum, vagus nerve, esophagogastric junction, proximal stomach, mid-stomach, distal antrum, hepatic artery, and left gastric artery, with the needle cap removed under direct vision throughout the procedure.

SUMMARY:
The goal of this clinical trial is to learn if combining Dexmedetomidine infusion and paragastric autonomic neural block will enhance the postoperative recovery of patients undergoing laparoscopic sleeve gastrectomy. The main questions it aims to answer are:

Will combining the two techniques (Dexmedetomidine infusion and paragastric autonomic neural block) improve the quality of recovery? Will opioid consumption postoperatively decrease after combining those two techniques? Will the patients be able to start mobilizing sooner after surgery? Will the patient encounter less incidence of nausea and vomiting?

Researchers will asses the quality of the patients' recovery by reviewing the Quality of recovery 40 (QoR 40) questionnaire filled by the patients, assessing hemodynamic parameters intra- and postoperatively, recording the opioids consumed by the patients in the postoperative period, recording the time to first mobilization of the patient, and recording the incidence of nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

1. ASA II-III
2. 18-60 years
3. BMI of 35-50 kg/m²

Exclusion Criteria:

1. Patients with chronic pain disorders
2. Patients using gabapentin, chronic opioid users
3. Patients on anticoagulant therapy
4. Patients with history of upper gastrointestinal system surgery
5. Patients with liver, kidney, cardiovascular diseases
6. Patients with allergy to dexmedetomidine or bupivacaine

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2025-06-06 (Estimated); Study Completion 2025-06-18 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction | Postoperative day 1
  Patient satisfaction will be measured using the QoR 40 questionnaire, filled by the patients (ranging from 40, which is extremely poor quality of recovery to 200, which is excellent quality of recovery)

SECONDARY OUTCOMES:
Baseline Demographics | preoperative
  Age, sex, body mass index (BMI), comorbidities will be recorded
Heart Rate | Heart rate will be recorded prior to induction, post-induction, after the loading dose of dexmedetomidine, 4 hours and 12 hours postoperatively.
  heart rate (beats/min) will be monitored continuously every 5 minutes and recorded prior to induction, post-induction, after the loading dose of dexmedetomidine, 4 hours, and 12 hours postoperatively.
Blood Pressure | Blood pressure will be recorded prior to induction, post-induction, after the loading dose of dexmedetomidine, 4 hours, and 12 hours postoperatively.
  blood pressure (mmHg) will be monitored continuously every 5 minutes and recorded prior to induction, post-induction, after the loading dose of dexmedetomidine, 4 hours, and 12 hours postoperatively.
Opioid consumption | at 4, 8, 12 hours postoperative
  Total opioids consumed by the patients will be recorded at 4, 8, 12 hours postoperative
Time to mobilize | Immediately postoperatively (in minutes)
  The time to first mobilization (in minutes) of the patient will be recorded
Incidence of nausea and vomiting | Postoperative day 1
  The incidence of nausea and vomiting postoperatively will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Main University Hospital, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No